CLINICAL TRIAL: NCT00826592
Title: Comparison of Video-based Versus Written Patient Education on Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 200816693-1
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Atopic Dermatitis; Atopic Eczema; Infantile Eczema; Hand Eczema
Keywords: patient education; dermatology patient education; atopic dermatitis; atopic dermatitis education; atopic eczema; infantile eczema; hand eczema
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-based education arm (Experimental): Subjects receiving the video-based educational material
  Interventions: Other: Patient Educational Materials
- Written education arm: (Active Comparator): Subjects receiving the written educational material
  Interventions: Other: Patient Educational Materials

INTERVENTIONS:
Other: Patient Educational Materials — In the experimental arm, the intervention is the video-based patient educational material on atopic dermatitis. In the active comparison arm (control arm), the comparison intervention is written patient educational material on atopic dermatitis.
  Other Names: Patient educational materials on atopic dermatitis

SUMMARY:
The purpose of this study is to compare the effect of video-based patient education with written instruction on subjects' knowledge of atopic dermatitis and their disease severity, measured by the Patient-oriented Eczema Measure (POEM), after viewing the educational materials.

DETAILED DESCRIPTION:
We plan to conduct a randomized, controlled trial comparing the effect of video-based patient education with written instruction on subjects' understanding of atopic dermatitis and their disease severity.

Subjects randomized to the video-based education arm will be instructed to watch a video on the classifications, aggravating factors, and treatment of atopic dermatitis. Subjects randomized to the written education arm will receive written information on the classifications, aggravating factors, and treatment of atopic dermatitis. The contents of the video and the written educational materials will be comparable.

At the end of the study period, 3 months later, subjects will be interviewed regarding their comprehension and attitude towards video-based and written education materials. Additionally, we will use the Patient-oriented Eczema Measure (POEM) questionnaire to assess the difference in subjects' disease severity between the 2 arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent, may be men or women.
* Able to adhere to the study visit schedule and other protocol requirements.
* Capable of giving informed consent.

Exclusion Criteria:

* Non-English speaking individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Subjects' disease severity measured by the patient-oriented eczema measure (POEM). | 3 months

SECONDARY OUTCOMES:
Subjects'comprehension and attitude towards video-based and written education materials. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: April Armstrong, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical